CLINICAL TRIAL: NCT05208073
Title: Effectiveness of Cosmetic Therapy on Self-esteem and Depression for Elderly Residents in Long-Term Care Institutions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Tsui-Wei Chien, Assistant Professor, National Taipei University of Nursing and Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: C110043
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Long-Term Care; Aged
Keywords: Elderly Residents; Long-Term Care Institution; Depression; Self-esteem; Cosmetic Therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The experimental group received 6-week cosmetic therapy.
  Interventions: Behavioral: Cosmetic therapy
- Control group (No Intervention): The control group maintains the institution's original daily routine care.

INTERVENTIONS:
Behavioral: Cosmetic therapy — The cosmetic therapy in this study is once a week, 60 minutes each section for a total of 6-week. Cosmetic therapy uses the teaching materials to teach the subjects skincare and makeup operation steps and use the 10-minute limb stretching to relax their minds before the activity, and then lead the research subjects to use cotton pads to apply lotion and lotion. , female subjects used powder, eyebrow pencil, and lipstick (or lip balm) to complete weekly different-themed activities and hairstyling, while men performed weekly different theme activities and hairstyling.
  Arms: Intervention group

SUMMARY:
Cosmetic therapy provides a psychological effect on the elderly, improving their self-confidence and social participation. This study was conducted to investigate the effectiveness of cosmetic therapy to enhance the self-esteem and reduce depression of elderly residents in long-term care institutions. We expect that a 6-week cosmetic therapy will improve the elderly's mental health, including depression and self-esteem.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 65 years old.
* Having been admitted to a long-term care institution (conservation type) for three months.
* Be able to communicate in Mandarin, Taiwanese and written languages.
* The total score of Mini-mental state examination (MMSE) is higher than 24 points.
* The muscle strength of the left or right hand is 4 points (inclusive) or above, and the maintenance and makeup procedures can be operated with one or both hands.
* After the researcher's explanation, the participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Under the age of 65.
* The applicant has been admitted to a long-term care institution (conservation type) for less than three months.
* Unable to communicate in Mandarin, Taiwanese and written language.
* Participated in cosmetic therapy.
* Diagnosed with mental illness (except depression), dementia and delirium.
* Currently taking antidepressant drugs.
* Currently receiving depression-related treatment.
* The maintenance and makeup steps cannot be operated with assistance.
* Failure to sign the research consent form.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Geriatric Depression Scale short-form (GDS-SF) | Pre-test before cosmetic therapy intervention and post-test at the end of six-week cosmetic therapy
  Geriatric Depression Scale short-form is a 15-item scale; each item on this scale uses a " Yes/ NO" answer method, and the scoring method is 1 point and 0 points. The total score ranges from 0 to 15, with less than 5 indicating no depression symptoms, 5 to 9 indicating mild depression, greater than or equal to 10 indicating moderate to severe depression.
Rosenberg Self-Esteem Scale (Chinese version) | Pre-test before cosmetic therapy intervention and post-test at the end of six-week cosmetic therapy
  Rosenberg Self-Esteem Scale (Chinese version) is a 10-item scale that measures the respondent's self-esteem. Each item is scored on a 4-point Likert scale, ranging from 1 (strongly disagree) to 4 (strongly agree); the minimum and maximum scores on the scale are 10 and 40, with lower scores suggesting better self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Tsui-Wei Chien, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Yi-xing Elderly long-term care center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No